CLINICAL TRIAL: NCT04762862
Title: QUANTACT : Impact of Pangenomic QUANTitative Alterations in Cancer Therapy
Acronym: QUANTACT
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 21LGTS01
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
"Precision medicine and targeted therapies have played a crucial role over the past ten years in the personalized care of cancer patients. In this retrospective and observational study, we focused on patients for which no standard or curative treatment was available and for which the management was discussed in a Molecular Tumor Board (MTB).

The role of the MTB is to decide the most appropriate therapeutic options for patients according to the potential identification of molecular targets.

Among the analyses carried out, we focused on a quantitative genome-wide analysis: the CGH/SNP-array (Comparative Genomic Hybridization / Single Nucleotide Polymorphism on array). The objective was to evaluate the impact of CGH/SNP-array analyses in the identification of targeted molecular alterations.

"

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor malignancy that is advanced or metastatic ;
* no standard or curative treatment available;
* non-opposition of the patient collected.

Exclusion Criteria:

* multiple cancer patient;
* ECOG Scale of Performance Status (PS) ≥2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients for which no standard or curative treatment was available and for which the personalized management was discussed in a Molecular Tumor Board.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of targeted molecular alterations | at day 0
  Number of targeted molecular alterations

SECONDARY OUTCOMES:
Number of patients eligible for targeted therapy (clinical trials or "off-label" drug) | at day 0
  Number of patients eligible for targeted therapy (clinical trials or "off-label" drug)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No